CLINICAL TRIAL: NCT04227769
Title: IL-1-receptor Antagonist During Cephalic Phase of Insulin Secretion in Health and Type 2 Diabetes
Acronym: Cephalira
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Too low recruitment in group with patients with diabetes.
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: EKNZ 2019-02307
Record Dates: First submitted 2020-01-07; First posted 2020-01-14 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus Type 2 in Obese; Inflammation; Metabolic Disease; Glucose Metabolism Disorders (Including Diabetes Mellitus)
Keywords: anakinra; cephalic phase of insulin secretion
MeSH Terms: conditions — Inflammation; Metabolic Diseases; Glucose Metabolism Disorders | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomized, double-blinded and open-label, placebo-controlled, partly cross-over clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- healthy individuals (Experimental): Two crossover visits with a washout period of at least 4 days in-between visits and at most two weeks: A) subcutaneous saline injection 3h before an oral standardized meal, B) subcutaneous injection of 100 mg of the IL-1 receptor antagonist anakinra 3h before an oral standardized meal. Treatments will be placebo controlled, crossover, double blinded. Standard dose of Anakinra (Kineret®; r-metHuIL-1ra, Swedish Orphan Biovitrum AB), i. e. 100 mg/ 0.67 ml s. c. or 0.67 ml of saline s. c. (placebo)
  Interventions: Drug: Anakinra Prefilled Syringe
- obese patients with type 2 diabetes (Experimental): Three crossover visits with a washout period of at least 4 days in-between: A) subcutaneous saline injection 3h before an oral standardized meal, B) subcutaneous injection of 100 mg of the IL-1 receptor antagonist anakinra 3h before an oral standardized meal, C) Additionally, after the second study day, participant in group 2 will be trained to self-inject the medication for 6 days. On the 7th day, an oral standardized meal test will be performed. Standard dose of Anakinra (Kineret®; r-metHuIL-1ra, Swedish Orphan Biovitrum AB), i. e. 100 mg/ 0.67 ml s. c. or 0.67 ml of saline s. c. (placebo)
  Interventions: Drug: Anakinra Prefilled Syringe

INTERVENTIONS:
Drug: Anakinra Prefilled Syringe — Subcutaneous injection of 100 mg/ 0.67 ml of Kineret or placebo
  Other Names: Kineret

SUMMARY:
A prospective, randomized, mixed double- and single-blinded, placebo-controlled, cross-over clinical trial to test whether acute treatment with an IL-1 receptor antagonist impacts insulin secretion over time during the cephalic phase, defined as the first 10 minutes after the first sensorial contact to food, in healthy individuals in healthy humans (Group 1) and in obese patients with type 2 diabetes (Group 2).

DETAILED DESCRIPTION:
The role of the immune system in metabolism has been extensively investigated in pancreatic islets and insulin sensitive tissues. However little attention has been given to a potential role of the innate immune system in the cephalic phase of insulin secretion. In humans, the cephalic phase of insulin secretion appear reduced in obesity and in patients with type 2 diabetes.

In this prospective, randomized, mixed double- and single-blinded, placebo-controlled, cross-over clinical trial we aim to test whether acute treatment with an IL-1 receptor antagonist impacts insulin secretion over time during the cephalic phase, defined as the first 10 minutes after the first sensorial contact to food, in healthy individuals in healthy humans (Group 1) and in obese patients with type 2 diabetes (Group 2).

Group 1: After screening, subjects will be randomized to two crossover visits with a washout period of at least 4 days in-between visits and at most two weeks: A) subcutaneous saline injection 3h before an oral standardized meal, B) subcutaneous injection of 100 mg of the IL-1 receptor antagonist anakinra 3h before an oral standardized meal. Treatments will be placebo controlled, crossover, double blinded. The study will be performed in a population of healthy individuals.

Group 2: Same as for Group 1 with the following addition: after the second study day, participant in group 2 will be trained to self-inject the medication for 6 days. On the 7th day, an oral standardized meal test will be performed.

Healthy subjects from group 1 will be matched for sex and age to the diabetic cohort from group 2.

ELIGIBILITY:
Inclusion criteria:

Main inclusion criteria:

* Age ≥ 18 years and ≤ 70 years at screening
* Male or female of non-child-bearing potential (meaning for women: not currently pregnant, post-menopausal female or using condoms and either intrauterine devices or 3-monthly contraceptive injection or birth-control pill.)

Healthy subjects:

* No apparent disease requiring medication
* BMI < 25 kg/ m2
* C-reactive protein ≤ 2 mg/L

Obese diabetic type 2 subjects:

* Type 2 diabetes
* HbA1c 7.0 -10.0%
* BMI ≥ 30.0 kg/m2
* C-reactive protein ≥ 2 mg/L

Exclusion criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Aversion or allergy to paracetamol or any component of the meal.
* Known history of allergy or hypersensitivity to any component of the investigational product formulations
* Concomitant treatment with GLP-1 agonists, DPP-4 inhibitors, insulin or insulin derivative
* Change in diabetes medication within the last 30 days
* Any biologic drugs targeting the immune system
* Fever, or other signs of infection requiring antibiotics within 3 weeks prior to screening, history of recurrent infection, immunodeficiency, known HIV or tuberculosis infection, active foot ulcer
* Participation in another study with investigational drug within 30 days prior to Screening and during the present study
* eGFR < 30 mL/min/1.73m2 per MDRD formula or kidney transplant (regardless of renal function)
* Known active or recurrent hepatic disorder (including cirrhosis, hepatitis B and hepatitis C, or confirmed ALAT/ASAT levels > 3 times ULN or total bilirubin > 2 times ULN),
* Haemoglobin <10.0 g/dL, white blood cell <3.0 x 103/mm3, platelet count <125 x 103/mm3
* Atrial fibrillation and/or a pacemaker

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Change in insulin concentration in blood during the cephalic phase of insulin secretion in healthy individuals | 10 minutes
  Insulin concentration in blood at 0, 3,6 and 10 minutes after ingestion of a standardized meal in healthy individuals.
Change in insulin concentration in blood during the cephalic phase of insulin secretion in obese patients with type 2 diabetes | 10 minutes
  Insulin concentration in blood at 0, 3, 6 and 10 minutes after ingestion of a standardized meal in healthy individuals in obese patients with type 2 diabetes.

SECONDARY OUTCOMES:
Change of C-peptide | 6 hours
  Plasma level of c-peptide before and after a standardized meal after acute treatment or repeated treatment with anakinra or placebo. Repeated Treatment applies only to anakinra and to Group 2.
Change of insulin | 6 hours
  Plasma level of insulin before and after a standardized meal after acute treatment or repeated treatment with anakinra or placebo. Repeated Treatment applies only to anakinra and to Group 2.
Change of glucose | 6 hours
  Plasma level of glucose before and after a standardized meal after acute treatment or repeated treatment with anakinra or placebo. Repeated Treatment applies only to anakinra and to Group 2.
Change of glucagon | 6 hours
  Plasma level of glucagon before and after a standardized meal after acute treatment or repeated treatment with anakinra or placebo. Repeated Treatment applies only to anakinra and to Group 2.
Change of GLP-1 | 6 hours
  Plasma level of GLP-1 before and after a standardized meal after acute treatment or repeated treatment with anakinra or placebo. Repeated Treatment applies only to anakinra and to Group 2.
Change of pancreatic polypeptide | 6 hours
  Plasma level of pancreatic polypeptide before and after a standardized meal after acute treatment or repeated treatment with anakinra or placebo. Repeated Treatment applies only to anakinra and to Group 2.
Change of IL-1β | 6 hours
  Plasma level of IL-1β before and after a standardized meal after acute treatment or repeated treatment with anakinra or placebo. Repeated Treatment applies only to anakinra and to Group 2.
Change of IL-6 | 6 hours
  Plasma level of IL-6 before and after a standardized meal after acute treatment or repeated treatment with anakinra or placebo. Repeated Treatment applies only to anakinra and to Group 2.
Change of IL-1Ra | 6 hours
  Plasma level of IL-1Ra before and after a meal through nasogastric tube or with anakinra or placebo after a standardized meal.
Change of TNFa | 6 hours
  Plasma level of TNFa before and after a standardized meal after acute treatment or repeated treatment with anakinra or placebo. Repeated Treatment applies only to anakinra and to Group 2.
change in hunger | 6 hours
  Visual analogue scale (VAS) for hunger (from minimum value = not hungry at all to maximum value = extremely hungry) before and after a standardized meal after acute treatment or repeated treatment with anakinra or placebo. Repeated Treatment applies only to anakinra and to Group 2.
Change in autonomic function | 6 hours
  Change in heart-rate variability during a continuous ECG as indirect measure of measure of the autonomic function before and after a standardized meal after acute treatment or repeated treatment with anakinra or placebo. Repeated Treatment applies only to anakinra and to Group 2.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Y Donath, Prof. Dr. MD, Principal Investigator — University of Basel
Locations (1):
- University Hospital Basel, Basel, Basel BS, Switzerland

IPD SHARING:
Plan to Share IPD: No